CLINICAL TRIAL: NCT05095909
Title: Utility of Intermittent Cryo-Compression Versus Traditional Icing Following Arthroscopic Rotator Cuff Repair
Acronym: ICC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICC2-2019
Record Dates: First submitted 2021-10-07; First posted 2021-10-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-09

CONDITIONS: Rotator Cuff Injuries; Cryotherapy Effect
Keywords: Cryo-compression; Rotator cuff repair
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cryo-compression (Experimental): Fitted with compression sleeve for the NICE Recovery SystemTM applied to the operative shoulder immediately post - operatively Minimum 6 hours treatment per day post-operatively. Utilize cyro-compression unit with a "Medium" compression level (inflate to 35 mmHg for 2 minutes and then deflate to 5 mmHg for 30 seconds) and "Level 3" cooling (50F (10C)) for the first 24 hours. After that time, the compression and cooling levels will be up to the patients' discretion.
  Interventions: Device: Cryo-compression
- Cryo-therapy (Active Comparator): Fitted with a standard gel ice pack with wrap immediately post-operatively. Minimum 6 hours treatment per day using gel ice packs.
  Interventions: Other: Cryo-therapy

INTERVENTIONS:
Device: Cryo-compression — Programmable intermittent compression with integrated cryo-therapy.
  Other Names: NICE Cold Therapy
  Arms: Cryo-compression
Other: Cryo-therapy — Subjects are fitted with gel ice packs and wraps.
  Other Names: Gel ice pack
  Arms: Cryo-therapy

SUMMARY:
Effective post - operative pain control following orthopedic surgical procedures without excessive reliance upon opioid pain medication has garnered increased attention in recent years. This study will evaluate the utilization of a non-invasive, novel cryo - compression, post-operative modality to improve pain control versus standard ice wraps in the immediate post-operative phase of arthroscopic rotator cuff surgery via a randomized controlled study design. Furthermore, if this study demonstrates improved pain control, improved quality of life and decreased opioid usage with the intermittent cold compression unit, recommendations may be considered for system-wide utilization.

DETAILED DESCRIPTION:
The purpose of this study is to test the proposed increase efficacy of combining both cold and compression modalities through cryo-compression therapy in post-operative pain management in arthroscopic rotator cuff repair surgery versus a control group of standard ice wraps. As opioid use within the field of orthopedics continues to grow as an area of investigation, surgeons must look elsewhere for pain management tactics.

Objectives of this study include:

1. Evaluate effectiveness of intermittent cryo-compression therapy versus standard ice wraps for post - operative pain control through patient reported visual analog pain scores and patient - reported opioid usage in patients undergoing arthroscopic rotator cuff repair.
2. Evaluate effectiveness of intermittent cryo-compression therapy versus standard ice wraps for reduction of post - operative tissue swelling in patients undergoing arthroscopic rotator cuff repair.
3. Determine cost comparison of intermittent compression cryotherapy versus interscalene catheter via historical controls as well as versus standard ice wraps.
4. Evaluate effect of intermittent cryo-compression therapy versus standard ice wraps on patient - reported quality of life via PROMIS.

Patients that are candidates for arthroscopic rotator cuff repair and complete informed consent process will be enrolled in study if no exclusion criteria are present. The study has determined an enrollment goal of 100 subjects (50 intermittent cryo-compression therapy, 50 standard cryo -therapy).

Following informed consent, patients enrolled in the study will be randomized in a 1:1 ratio using permuted blocks of sizes 2 and 4 to have post-operative cryotherapy using ice packs or with the intermittent cold compression therapy unit. Randomization assignments will be contained in sequentially numbered, opaque, sealed envelopes, which will be prepared by an individual not involved in patient consent or patient treatment. After the patient is consented, the next envelope in the sequence will be opened and the patient will be assigned to a group following the treatment listed in the envelope.

Prior to surgery, the subject will complete pre-operative data collection. The subject will be given a tracking diary in order to record immediate post-operative data through the first post-operative visit. Subjects will undergo arthroscopic rotator cuff repair by a single surgeon as a standard of care procedure.

Subjects randomized to the study group will have the compression sleeve for the NICE Recovery SystemTM applied to the operative shoulder immediately post - operatively and those randomized to the control group a standard gel ice pack with wrap. Each will use the assigned version of cold therapy with a goal of 6 hours daily and will record overages using one half hour as a minimum unit.

After enrollment and surgery, subjects will follow a post-operative follow-up visit schedule including 2-days, first post-operative visit, 60 days, 3 months, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are candidates for arthroscopic rotator cuff repair

   1. Acute, traumatic tear of the rotator cuff in an active patient
   2. Chronic, symptomatic tear of the rotator cuff in an active patient having failed non - operative treatment
2. Patient agreeable to participation in the study and able to complete informed consent process and all study requirements.
3. ≥18 years of age

Exclusion Criteria:

1. Pregnancy (per pre-operative physical)
2. Presence of significant glenohumeral joint osteoarthritis
3. Age over 70
4. History of clinically diagnosed lymphedema
5. Morbid obesity (BMI > 45)
6. History of drug or alcohol addiction, prior opioid dependence, or current use of opioid medication (preoperative)
7. Investigators concern regarding subject's ability or willingness to follow protocol.
8. History of significant vascular impairment in the affected region (e.g., from prior frostbite, diabetes, arteriosclerosis or ischemia).
9. History of acute paroxysmal cold hemoglobinuria or cryoglobulinemia.
10. History of Raynaud's disease or cold hypersensitivity (cold urticarial).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pain levels in the post-operative period using VAS Pain Scale. | up to 15 days
  Evaluate effectiveness of intermittent cryo-compression therapy versus standard ice wraps for post - operative pain control through patient reported visual analog pain scores and patient - reported opioid usage in patients undergoing arthroscopic rotator cuff repair. Pain levels will be documented by the VAS Pain Scale
Evaluation of post-operative edema comparing pre-operative and post-operative upper arm measurements. | up to 15 days
  Evaluate effectiveness of intermittent cryo-compression therapy versus standard ice wraps for reduction of post - operative tissue swelling in patients undergoing arthroscopic rotator cuff repair by measuring circumference (inches) of upper arm using a flexible measuring tape.

SECONDARY OUTCOMES:
Cost analysis of post-operative cryotherapy modalities and other historical controls of pain post-operative pain control. | 10 days
  Determine cost differential of intermittent compression cryotherapy versus interscalene catheter via historical controls as well as versus standard ice wraps.
Quality of life evaluation comparison of post-operative cryotherapy modalities using PROMIS Global-10 scale. | 1 year
  Evaluate effect of intermittent cryo-compression therapy versus standard ice wraps on patient - reported quality of life via Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10

CONTACTS AND LOCATIONS:
Overall Officials: L Pearce McCarty III, MD, Principal Investigator — Allina Health
Locations (1):
- Allina Health Orthopedics, Plymouth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No